CLINICAL TRIAL: NCT04396782
Title: Effectiveness of Immersive Virtual Reality in Functional Rehabilitation in Older People With Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Collaborators: Carmen Ruiz Vergara (Unknown); Rocío Martín Valero (Unknown)
Responsible Party: Principal Investigator, Rocío Martín Valero, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UMALAGARV Knee
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physiotherapy rehabilitation with IVR (Experimental): This program includes: static bicycle with virtual reality glasses, analytical lower limb exercises, global lower limb exerciseswith virtual reality glasses and activities to be done at home.
  Interventions: Other: standard physiotherapy rehabilitation
- standard physiotherapy rehabilitation (Active Comparator): static bicycle, analytical lower limb exercises, global lower limb exercises and activities to be done at home.
  Interventions: Other: Physioterapy rehabilitation with IVR

INTERVENTIONS:
Other: Physioterapy rehabilitation with IVR — This program includes: static bicycle with virtual reality glasses, analytical lower limb exercises, global lower limb exerciseswith virtual reality glasses and activities to be done at home.
  Arms: standard physiotherapy rehabilitation
Other: standard physiotherapy rehabilitation — static bicycle, analytical lower limb exercises, global lower limb exercises and activities to be done at home.
  This group will perform only five minutes of virtual reality play, but will not use their lower limbs. This way, the results of rehabilitation will not be affected and therapists and patients will be blinded.
  Arms: physiotherapy rehabilitation with IVR

SUMMARY:
The number of knee arthroplasties performed each year is constantly increasing. Although the outcome is generally favourable, 10-20% do not achieve a satisfactory clinical result. This study evaluates the effectiveness of immersive virtual reality rehabilitation in older people who have undergone knee arthroplasty surgery. The 6 Meter Walking Test is used to determine the improvement of patients after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* people who are admitted to one of the two chosen residences on the Costa del Sol who have had, or will have, a total knee arthroplasty recently.
* People between 60-75, who want to receive rehabilitation treatment.

Exclusion Criteria:

* Patients who refuse to participate or who suffer serious post-operative complications.
* patients with neurological or cognitive impairment that could interfere with the performance of the rehabilitative treatment will be excluded.
* Those with any severe cardiovascular or pulmonary disease that would prevent them from exercising and also those who are not allowed physical activity for any reason.
* Those with poor visual acuity who are unable to see the visual characteristics of the screen.
* Patients with severe contralateral knee osteoarthritis (>5/10 pain when climbing stairs) or other orthopaedic conditions that limited function and required an alternative simultaneous operation, e.g. severe lumbar spinal stenosis, severe OA of the hip or ankle...
* Those who are scheduled for other lower limb surgery in the next 6 months.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in six meter walking test (6-MWT) score | Baseline, up to three an six months.
  Six-meter walking test is a a well-established outcome measure in a variety of diseases. It is accurate, reproducible, simple to administer, and well tolerated. The 6MWT is a robust assessment tool for use in clinical trials given its ability to quantitatively evaluate ambulation in a controlled environment.
  Participants will be asked to do quick laps in a flat corridor for 6 minutes with the verbal stimulus provided by the assessor at the end of each lap.
  A significant improvement threshold after surgery could be between 26 and 55m

SECONDARY OUTCOMES:
Sit to Stand Test | Baseline, up to three an six months.
  Sit to Stand Test is a simple test to evaluate lower limb muscle strength and balance ability. This test measures the time it takes to sit down completely and get up 5 times with arms crossed over the chest and using a standard height chair (46cm).
The range of motion | Baseline, up to three an six months.
  The range of motion (ROM) of knee flexion and extension measured with a goniometer.
The Oxford Knee Score (OKS) | Baseline, up to three an six months.
  The Oxford Knee Score (OKS) is a specific measurement for assessing knee function and condition.
  It consists of 12 patient-reported questions that measure pain and function after knee arthroplasty surgery. Each question is scored from 0 to 4 with 4 being the best result, producing overall scores that range from 0 to 48, 48 being the best result.
The BERG scale | Baseline, up to three an six months.
  The BERG scale which is a valid and sensitive scale for assessing balance in the elderly.
  It is based on the performance of 14 common balance tasks, experienced in daily life, which are graded on an ordinal scale of 5 points (0-4) with a maximum score of 56.
  Higher scores indicate better balance.
The McMaster Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, up to three an six months.
  The McMaster Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) is a specific questionnaire to assess the treatment effects of osteoarthritis on patients and their health-related quality of life.
  It is composed of a multidimensional scale with 24 items grouped in three dimensions: pain (5 items), stiffness (2 items) and physical function (17 items). They are answered by a Likert-type scale with 5 levels of response representing different degrees of intensity (none, mild, moderate, severe, extreme) scoring from 0 to 4. The final score is the sum of the scores of each item. The higher the score, the worse the patient's condition. The data are standardized on a range of 0 (best health condition) to 100 (worst possible condition).
The User Satisfaction Evaluation Questionnaire | up to six months
  The User Satisfaction Evaluation Questionnaire (USEQ) is a questionnaire to evaluate the satisfaction and ease of use of virtual rehabilitation systems.
  It includes, with a 5-point Likert scale, 6 questions which we can see in Annex 4. The total score ranges from 6 (low satisfaction) to 30 (excellent satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No